CLINICAL TRIAL: NCT07258095
Title: INNOV5-MH-MAROC: Multicenter Pragmatic Randomized Controlled Trial Evaluating an Integrated Program of Five WHO Innovations in Mental Health in Morocco
Brief Title: INNOV5-MH-MAROC: Integrated Mental Health Care for Adolescents and Adults in Primary Care Centers and Schools in Morocco
Acronym: INNOV5-MH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Medical Academy Maroc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMA-INNOV5-MH-MAROC-01; SMA-INNOV5-MH-MAROC-01 (Other: Swiss Medical Academy Maroc)
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Depression in Adolescence; Depression in Adults; Anxiety; Mental and Behavioural Disorders
Keywords: Depression; Anxiety; Adolescent mental health; Primary care; School-based mental health; Digital mental health; Virtual reality exposure; mhGAP; Task-shifting; Morocco
MeSH Terms: conditions — Anxiety Disorders; Mental Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Participants are randomized 1:1 to either the INNOV5 integrated mental health program or enhanced treatment as usual (TAU+) in a two-arm parallel-group pragmatic trial conducted in Moroccan primary care centers and high schools.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INNOV5 Integrated Program (Experimental): Participants receive the INNOV5 integrated mental health program combining: (1) a collaborative care model in primary care; (2) mhGAP-based task-shifting and stepped care; (3) validated digital mental health interventions (apps and online tools); (4) virtual reality exposure therapy for selected anxiety- or trauma-related cases; and (5) a school-based mental health promotion component in participating high schools.
  Interventions: Behavioral: INNOV5 Integrated Mental Health Program; Behavioral: Enhanced Treatment as Usual (TAU+)
- Enhanced Treatment as Usual (TAU+) (Active Comparator): Participants receive enhanced treatment as usual in participating primary care centers and schools. TAU+ consists of routine mental health care and referrals available at each site, plus minimal enhancements such as access to WHO mhGAP materials and basic information and referral resources. Participants do not receive the specific INNOV5 program components.
  Interventions: Behavioral: INNOV5 Integrated Mental Health Program; Behavioral: Enhanced Treatment as Usual (TAU+)

INTERVENTIONS:
Behavioral: INNOV5 Integrated Mental Health Program — Integrated multicomponent mental health program combining: (1) a collaborative care model in primary care; (2) mhGAP-based task-shifting and stepped care; (3) validated digital mental health interventions (apps and online tools); (4) virtual reality exposure therapy for selected anxiety- or trauma-related cases; and (5) a school-based mental health promotion component in participating high schools.
Behavioral: Enhanced Treatment as Usual (TAU+) — Usual mental health care and referrals available at participating primary care centers and schools, with minimal enhancements such as WHO mhGAP materials and basic information and referral resources, but without access to the INNOV5 integrated program components.

SUMMARY:
Depression and anxiety are highly prevalent among adolescents and adults in Morocco, while access to evidence-based care in primary care centers and schools remains limited. This multicenter pragmatic randomized controlled trial evaluates an integrated mental health program inspired by WHO priorities. The INNOV5 intervention combines: (1) a collaborative care model in primary care; (2) mhGAP-based task-shifting and stepped care; (3) validated digital mental health interventions; (4) virtual reality exposure therapy for selected anxiety- or trauma-related cases; and (5) a school-based mental health promotion component in participating high schools. The primary objective is to compare the change in depressive symptoms (PHQ-9) at 6 months between INNOV5 and enhanced treatment as usual (TAU+). Secondary objectives include effects on anxiety (GAD-7), quality of life (WHOQOL-BREF), suicidal ideation and behavior (C-SSRS), functioning, school attendance, and feasibility and acceptability of the program.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents (12-17 years) and adults (≥18 years) attending participating primary care centres or high schools in Morocco.
* Clinically significant depressive and/or anxiety symptoms identified by screening (PHQ-9 and/or GAD-7) according to study thresholds.
* Able to understand study procedures and provide informed consent (or parental consent and adolescent assent for minors).
* Planning to remain in the study area for at least 12 months.

Exclusion Criteria:

* Acute psychiatric emergency requiring immediate specialised care (e.g. psychosis, high-risk suicidal crisis, severe substance use disorder).
* Cognitive impairment or severe medical condition preventing participation in the intervention or assessments.
* Current participation in another interventional mental health trial.
* Any other situation judged by the investigator to make participation unsafe or inappropriate.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2028-03-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in depressive symptoms (PHQ-9) | Baseline to 6 months
  Mean change in Patient Health Questionnaire-9 (PHQ-9) total score from baseline to 6 months comparing INNOV5 versus enhanced treatment as usual (TAU+). The PHQ-9 is a 9-item self-report scale of depressive symptoms; total scores range from 0 to 27, with higher scores indicating more severe depressive symptoms.

SECONDARY OUTCOMES:
Change in anxiety symptoms (GAD-7) | Baseline to 6 months
  Mean change in Generalized Anxiety Disorder-7 (GAD-7) total score from baseline to 6 months between participants allocated to the INNOV5 integrated mental health program and those allocated to enhanced treatment as usual (TAU+). The GAD-7 is a 7-item self-report measure of anxiety symptoms; total scores range from 0 to 21, with higher scores indicating more severe anxiety.

OTHER OUTCOMES:
Change in quality of life (WHOQOL-BREF) | Baseline to 6 months
  Change in health-related quality of life measured by the WHOQOL-BREF. The WHOQOL-BREF is a 26-item self-report questionnaire assessing four domains (physical health, psychological health, social relationships and environment). Domain scores are transformed to a 0-100 scale, with higher scores indicating better quality of life. Mean change in WHOQOL-BREF domain scores from baseline to 6 months will be compared between participants allocated to the INNOV5 integrated mental health program and those allocated to enhanced treatment as usual (TAU+).

CONTACTS AND LOCATIONS:
Locations (1):
- Swiss Medical Academy Maroc, Sion, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the primary and secondary outcome analyses will be made available to qualified researchers upon reasonable request, after completion of the trial and publication of the main results. Data sharing will comply with Moroccan data protection law (Loi 09-08), CNDP authorization and institutional policies. A data sharing agreement will be required.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From 12 months after publication of the primary trial results and for up to 5 years thereafter.
Access Criteria: Researchers must submit a brief research proposal and analysis plan to the Swiss Medical Academy data access committee (contact@swissmedicalacademy.ma
  ). Requests will be reviewed for scientific merit, ethical approval and compliance with data protection regulations. Upon approval and signature of a data sharing agreement, de-identified IPD will be transferred via a secure data sharing platform.